CLINICAL TRIAL: NCT06576310
Title: Evaluation of Predictive Factors for Dental Occlusal Changes in the Treatment of Obstructive Sleep Apnea With Mandibular Advancement Appliance
Brief Title: Predictive Factors for Occlusal Changes in Obstructive Sleep Apnea Treatment With Mandibular Advancement Appliance
Acronym: APNEAMOUVE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0024
Record Dates: First submitted 2024-08-01; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: MAD therapy; side effect; Dental occlusion; electromyography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Bites and Stings | interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA patients with mandibular advancement appliance: Patients with obstructive sleep apnea (OSA) treated with a mandibular advancement device (MAD), monitored for changes in masticatory muscle activity and occlusal modifications over a 6-month period. The study involves routine clinical visits and additional assessments including electromyography (EMG) with and without the appliance, optical impressions, digital occlusion recordings, patient diaries, and questionnaires on quality of life, temporo mandibular dysfunction pain, oral habits, stress and anxiety, and sleep evaluation.
  Interventions: Device: Mandibular Advancement Device

INTERVENTIONS:
Device: Mandibular Advancement Device — In this research, participation in the protocol seamlessly integrates into routine care at the Odontology Department of the University Hospital of Toulouse. The visits include the provision of the orthosis at 3 weeks (T1), with EMGs and digital occlusal analysis. The 6-week follow-up visit (T2) adjusts therapeutic propulsion, subjectively resolving symptoms related to OSAS. At the T0 visit, the researchers collect the polysomnographic monitoring before fitting the orthosis (carried out in the patient's reference sleep laboratory) to assess treatment efficiency. The end-of-research visit (6 months after T1) comprehensively collects data, including questionnaires on stress, anxiety, sleep quality and quantity, oral habits, temporo mandibular dysfunction pain, and quality of life. Moreover, the researchers collect the polysomnographic monitoring after 3 months fitting the orthosis (carried out in the same patient's reference sleep laboratory than before fitting the orthosis).

SUMMARY:
This research addresses obstructive sleep apnea syndrome (OSAS), affecting 6-12% of French adults, often treated with mandibular advancement devices (MADs). MADs may lead to occlusal modifications, causing a 50% treatment abandonment rate. The study employs surface electromyography to assess masticatory muscle activity before and during MAD use, correlating it with occlusal changes after 6 months. The primary goal is to determine dental displacement profiles post-6-month MAD treatment, providing insights for personalized care and minimizing treatment failures.

DETAILED DESCRIPTION:
In this exploratory electro-pathophysiological study, our objective is to provide a significant contribution to understanding the underlying mechanisms of occlusal modifications associated with mandibular advancement device (MAD) treatment in patients suffering from obstructive sleep apnea syndrome (OSAS). Drawing from observational data, the researchers aim to identify specific electrophysiological profiles linked to masticatory muscle activity, correlating with occlusal changes after MAD treatment. This innovative approach involves detailed data collection on electrophysiological profiles, initial clinical characteristics pre-treatment, and post-treatment follow-up data. Focusing on patients from the dentistry department at Toulouse University Hospital, the study seeks to establish correlations between muscle activity recorded before and during MAD treatment and occlusal changes, ultimately defining electrophysiological patient profiles. These profiles could potentially guide personalized care, anticipating risks of occlusal modifications and reducing treatment dropouts or failures.

The study utilizes diverse exams-orthopantomogram, optical impressions, surface electromyography, polysomnography, and research questionnaires. Data collected pre- and post-mandibular advancement device treatment for six months will innovatively analyze the links between masticatory muscle activity and occlusal changes, aiming to define specific electrophysiological patient profiles.

In this research, participation in the protocol seamlessly integrates into routine care at the Odontology Department of the Toulouse University Hospital. The visits include the provision of the orthosis at 3 weeks (T1), with EMGs and digital occlusal analysis. The 6-week follow-up visit (T2) adjusts therapeutic propulsion, subjectively resolving symptoms related to OSAS. At the T0 visit, the researchers collect the polysomnographic monitoring before fitting the orthosis (carried out in the patient's reference sleep laboratory) to assess treatment efficiency.(The end-of-research visit (6 months after T0) comprehensively collects data, including questionnaires on stress, anxiety, sleep quality and quantity, oral habits, temporo mandibular dysfunction pain, and quality of life. Moreover, the researchers collect the polysomnographic monitoring after 3 months fitting the orthosis (carried out in the same patient's reference sleep laboratory than before fitting the orthosis).

ELIGIBILITY:
Inclusion Criteria:

* Patient with complete dentition (up to second molars)
* Polysomnography or polygraphy
* Diagnosis of OSA
* Patient receiving OAM treatment at the Odontology Department of Toulouse University Hospital
* Patient with contemporary panoramic and lateral cephalometric X-rays (common practice) taken at the time of orthotic treatment
* Individual affiliated with or covered by a social security scheme
* Voluntary, informed, written consent, signed by both participant and investigator (prior to inclusion and any necessary research-related examinations).

Exclusion Criteria:

* Inability to provide informed consent
* Pregnant or breastfeeding patient
* Patient with curators, guardians, or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with sleep apnea treated with a mandibular advancement device
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
OCCLUSAL MODIFICATIONS AFTER 6 MONTHS OF OAM TREATMENT | 6 month
  assessment of occlusal modifications after 6 months of mandibular advancement device (OAM) treatment. Dental occlusion will be measured using digital occlusal analysis with OCCLUSENS® (Bausch; Köln, Germany), considering the extent of contacts (centroid) and their intensity (%), and through morphometric analysis based on optical impressions obtained pre and post-treatment using the TRIOS optical camera (3Shape, Dentsply®)
PRIMARY EXPOSURE VARIABLE: MASTICATORY MUSCLE ACTIVITY | 6 month
  The primary exposure of interest is the activity of masticatory muscles measured by EMG, in the form of motor-evoked potentials (MEPs in µV/s). This measurement will be conducted at the T1 visit when the orthosis is provided to the patient (3 weeks after inclusion) and 6 months after the inclusion visit. At each measurement time, surface EMG will be conducted bilaterally (4 locations in total), both with and without OAM. The association between muscle activity at inclusion and occlusal modifications will be studied for the primary objective, while the association between muscle activity after 6 months of treatment and occlusal modifications will be explored as a secondary objective.

OTHER OUTCOMES:
OSA phenotype at T0 visit | baseline
  The phenotype is classified as:
  * Typical OSA with somnolence,
  * Female OSA with insomnia, depression, and a relatively strong association with arterial hypertension and metabolic comorbidities,
  * OSA in elderly subjects with comorbidities,
  * OSA in young subjects with predominantly nocturnal respiratory symptoms and minimal daytime disturbance.
initial sleep assesment | baseline
  Sleep will be assessed with polysomnography Oxygen desaturation index A normal oxygen saturation level should be about 96 to 97%. When blood oxygen levels drop below 90% Oxygen Desaturation Index is considered slightly abnormal. When blood oxygen levels dip even lower to 80 or 89%, they are considered moderately abnormal. Any blood oxygen levels below 80% are considered severe.
Therapeutic mandibular advancement assessed at the T2 visit | 6 weeks
  As a percentage of voluntary mandibular protrusion and in mm of advancement
Titration modality assessed at the T2 visit | 6 weeks
  Conventional and with a medical titration aid device
difference in Patient's clinical characteristics at 6 months | 6 months
  Difference in :
  - Body Mass Index (BMI),
Clinical characteristics | 6 months
  - Duration of MAD wear,
Clinical characteristics | 6 months
  - Frequency of MAD wear.
Patient's quality of life | baseline
  Measured by the Short Form Survey (SF-36)
Patient's quality of life | 6 months
  Measured by the SF-36 questionnaire. Scoring the 36-Item Health Survey is a two-step process. First, all items are scored so that a high score defines a more favorable health state.
  In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
  In step 2, items in the same scale are averaged together to create the 8 scale scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores.
  Hence, scale scores represent the average for all items in the scale that the respondent answered.

CONTACTS AND LOCATIONS:
Overall Officials: Constance CUNY, MD, Principal Investigator — University Hospital, Toulouse